CLINICAL TRIAL: NCT05795179
Title: Neural and Affective Mechanisms Underlying Prospective Self-control Costs
Brief Title: Stress & Self-Control Costs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 22-01630
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Self-Control
MeSH Terms: conditions — Self-Control | interventions — Psychological Tests; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Physiological Stress (Experimental): Healthy dieters will undergo a single-visit neuroimaging study where they will first complete demographic and self-report measures followed by a self-control decision task in an fMRI scanner. Prior to scanning, participants will be assigned to a physiological stress group and complete the corresponding stress task. For the physiological stress group, this task is the Cold-Pressor Task (CPT), a physiological stress task in which participants continuously submerge their hand and forearm in ice-water (0-4°C) for 3 minutes. After the scan, participants will wait for 1 hour in an adjacent study room where they will play out one trial of the decision-making task completed in the scanner.
  Interventions: Behavioral: Cold-Pressor Task (CPT); Device: Functional Magnetic Resonance Imaging (fMRI)
- Social Stress (Experimental): Healthy dieters will undergo a single-visit neuroimaging study where they will first complete demographic and self-report measures followed by a self-control decision task in an fMRI scanner. Prior to scanning, participants will be assigned to the social stress group and complete the corresponding stress task. For the social stress group, this task is the Trier Social Stress Test (TSST), a psychosocial stressor that requires participants perform a short speech and solve math problems in front of 2 evaluative judges. After the scan, participants will wait for 1 hour in an adjacent study room where they will play out one trial of the decision-making task completed in the scanner.
  Interventions: Behavioral: Trier Social Stress Test (TSST); Device: Functional Magnetic Resonance Imaging (fMRI)
- Physiological Non-Stress (Active Comparator): Healthy dieters will undergo a single-visit neuroimaging study where they will first complete demographic and self-report measures followed by a self-control decision task in an fMRI scanner. Prior to scanning, participants will be assigned to the physiological non-stress group and complete the corresponding stress task. For the physiological non-stress group, participants will continuously submerge their hand and forearm in warm water for 3 minutes. After the scan, participants will wait for 1 hour in an adjacent study room where they will play out one trial of the decision-making task completed in the scanner.
  Interventions: Behavioral: Modified Non-Stress CPT; Device: Functional Magnetic Resonance Imaging (fMRI)
- Social Non-Stress (Active Comparator): Healthy dieters will undergo a single-visit neuroimaging study where they will first complete demographic and self-report measures followed by a self-control decision task in an fMRI scanner. Prior to scanning, participants will be assigned to the social stress group and complete the corresponding stress task. For the social non-stress group, participants will be asked to prepare for a speech that they will practice alone to themselves and complete math problems alone on a piece of scrap paper. After the scan, participants will wait for 1 hour in an adjacent study room where they will play out one trial of the decision-making task completed in the scanner.
  Interventions: Behavioral: Modified Non-Stress TSST; Device: Functional Magnetic Resonance Imaging (fMRI)

INTERVENTIONS:
Behavioral: Cold-Pressor Task (CPT) — CPT is a physiological stress task in which participants continuously submerge their hand and forearm in ice-water (0-4°C) for 3 minutes.
  Arms: Physiological Stress
Behavioral: Trier Social Stress Test (TSST) — The TSST is a psychosocial stressor that requires participants perform a short speech and solve math problems in front of 2 evaluative judges.
  Arms: Social Stress
Behavioral: Modified Non-Stress CPT — The modified non-stress CPT involves participants continuously submerging their hand and forearm in warm water for 3 minutes.
  Arms: Physiological Non-Stress
Behavioral: Modified Non-Stress TSST — For the modified non-stress TSST, participants are asked to prepare for a speech that they will practice alone to themselves and complete math problems alone on a piece of scrap paper.
  Arms: Social Non-Stress
Device: Functional Magnetic Resonance Imaging (fMRI) — Participants will complete the self-control task in the fMRI scanner.

SUMMARY:
Self-control failures are a universal challenge for healthy and clinical populations. Recent work suggests these failures may arise from excessive cognitive costs associated with exercising self-control, yet the mechanisms underlying these costs are unknown. To address this, the investigators will use a validated decision-making task that measures how much individuals will pay (from a study endowment) to restrict access to tempting rewards that may lead to self-control failures. The investigators will examine these costs to identify their cognitive, neural and affective mechanisms. First, the investigators will identify the cognitive and computational mechanism that gives rise to self-control costs. Second, the investigators will characterize the neural correlates of self-control costs and identify neural mediators and connectivity patterns stemming from these costs. Finally, the investigators will examine how different classes of stressors (physical, social, or lifetime stress) shape the behavioral and neural representations of self-control costs.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age, able to speak, read, and write fluently in English
* be willing and able to follow study procedures and provide informed consent.
* Must additionally confirm they are on a diet to maintain/lose weight and are implementing/maintaining dietary changes.

Exclusion Criteria:

* History of or medication for neurologic or psychiatric disease
* High-blood pressure or heart condition
* Diabetes, food allergies, metabolic disorders or history of eating disorder
* Use of corticosteroids or beta-blockers
* Metallic implants or devices contraindicating magnetic resonance imaging.
* Pregnancy is considered an exclusion criteria due to all stress and scanning procedures, thus pregnant participants will not be permitted to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Average Self-Control Cost | Day 1
  The self-control cost is the amount that a participant would be willing to pay to avoid temptation. This will be tested in a self-control task in which participants are shown an images of snack food and report how much they would be willing to avoid the different food items.
Change in fMRI BOLD Signal During Self-Control Decisions | Day 1 (Up to 1.5 Hours)
  Functional MRI (fMRI) data will be analyzed to measure changes in blood-oxygen-level-dependent (BOLD) signal in the Dorsal Anterior Cingulate Cortex (dACC), Frontopolar Cortex (FPC) and Orbitofrontal Cortex (OFC) regions of interest as participants make self-control cost decisions during the self-control activity.

CONTACTS AND LOCATIONS:
Overall Officials: Candace Raio, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: candace.raio@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to candace.raio@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.